CLINICAL TRIAL: NCT00305773
Title: A Phase 2 Study of Suberoylanilide Hydroxamic Acid (SAHA) in Acute Myeloid Leukemia (AML)
Brief Title: Vorinostat in Treating Patients With Acute Myeloid Leukemia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-01470; NCI-2012-01470 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CDR0000465213; JHOC-J0557; MAYO-MC0483; JHOC-J0550; NCI-6882; MC0483 (Other: Mayo Clinic); 6882 (Other: CTEP); N01CM62205 (NIH); P30CA015083 (NIH)
Record Dates: First submitted 2006-03-21; First posted 2006-03-22 (Estimated); Results first posted 2013-05-16 (Estimated); Last update posted 2014-05-19 (Estimated); Status verified 2012-12

CONDITIONS: Adult Acute Erythroid Leukemia (M6); Adult Acute Megakaryoblastic Leukemia (M7); Adult Acute Minimally Differentiated Myeloid Leukemia (M0); Adult Acute Monoblastic Leukemia (M5a); Adult Acute Monocytic Leukemia (M5b); Adult Acute Myeloblastic Leukemia With Maturation (M2); Adult Acute Myeloblastic Leukemia Without Maturation (M1); Adult Acute Myeloid Leukemia With 11q23 (MLL) Abnormalities; Adult Acute Myeloid Leukemia With Inv(16)(p13;q22); Adult Acute Myeloid Leukemia With t(15;17)(q22;q12); Adult Acute Myeloid Leukemia With t(16;16)(p13;q22); Adult Acute Myeloid Leukemia With t(8;21)(q22;q22); Adult Acute Myelomonocytic Leukemia (M4); Adult Acute Promyelocytic Leukemia (M3); Recurrent Adult Acute Myeloid Leukemia; Refractory Cytopenia With Multilineage Dysplasia; Secondary Acute Myeloid Leukemia; Untreated Adult Acute Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Erythroblastic, Acute; Leukemia, Megakaryoblastic, Acute; Leukemia, Monocytic, Acute; Leukemia, Myeloid, Acute; Congenital Abnormalities; Leukemia, Myelomonocytic, Acute; Leukemia, Promyelocytic, Acute | interventions — Vorinostat

ARMS (2):
- Arm I (once daily vorinostat) (Experimental): Patients receive oral vorinostat (SAHA) once a day on days 1-21. In both arms, treatment repeats every 21 days for up to 17 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: vorinostat
- Arm II (thrice daily vorinostat) (Experimental): Patients receive oral SAHA three times a day on days 1-14. In both arms, treatment repeats every 21 days for up to 17 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: vorinostat

INTERVENTIONS:
Drug: vorinostat — Given orally once daily
  Other Names: L-001079038; SAHA; suberoylanilide hydroxamic acid; Zolinza
  Arms: Arm I (once daily vorinostat)
Drug: vorinostat — Given orally three times daily
  Other Names: L-001079038; SAHA; suberoylanilide hydroxamic acid; Zolinza
  Arms: Arm II (thrice daily vorinostat)

SUMMARY:
Vorinostat may stop the growth of cancer cells by blocking some of the enzymes needed for their growth. Giving the drug in different ways may kill more cancer cells. This randomized phase II trial is studying two different schedules of vorinostat to see how well they work in treating patients with acute myeloid leukemia.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine the toxicity and the proportion of complete remissions associated with two different treatment schedules of vorinostat (SAHA) in patients with acute myeloid leukemia.

SECONDARY OBJECTIVES:

I. Determine the toxic effects of SAHA in this study population. II. Examine for preliminary evidence of re-expression of silenced genes in leukemic blasts in response to SAHA.

OUTLINE: This is a multicenter, randomized study. Patients are stratified according to disease status (relapsed vs untreated). Patients are randomized to 1 of 2 treatment arms.

ARM I: Patients receive oral vorinostat (SAHA) once a day on days 1-21. In both arms, treatment repeats every 21 days for up to 17 courses in the absence of disease progression or unacceptable toxicity.

ARM II: Patients receive oral SAHA three times a day on days 1-14. In both arms, treatment repeats every 21 days for up to 17 courses in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed periodically for up to 2 years.

PROJECTED ACCRUAL: A total of 44 patients will be accrued for this study.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of acute myeloid leukemia (AML), meeting 1 of the following criteria:

  * Relapsed AML in the following categories:

    * Good-risk cytogenetics [inv(16), t (8;21)] in second relapse or in first relapse following a remission of < 12 months
    * Acute promyelocytic leukemia (M3) in second relapse or greater AND must have relapsed following both tretinoin-anthracycline-based therapy and arsenic trioxide-based therapy
    * All other relapsed patients are eligible
  * Untreated AML in the following categories:

    * At least 65 years of age
    * Myelodysplastic syndromes-AML (AML with trilineage dysplasia)
    * AML with del5Q or monosomy 5, monosomy 7, or complex cytogenetics (≥ 3 cytogenetic abnormalities)
* Refused or ineligible for potentially curative options such as allogeneic stem cell transplantation
* No clinical evidence of CNS or pulmonary leukostasis, disseminated intravascular coagulation, or CNS leukemia
* ECOG performance status (PS) 0-2 or Karnofsky PS ≥ 60%
* Life expectancy ≥ 3 months
* Bilirubin normal unless attributed to hemolysis or Gilbert's disease in the opinion of the investigator
* AST/ALT ≤ 2.5 times upper limit of normal (ULN)
* Creatinine normal OR creatinine clearance ≥ 60 mL/min
* No history of allergic reactions attributed to compounds of similar chemical or biologic composition to vorinostat
* No uncontrolled intercurrent illness, including any of the following:

  * Ongoing or active infection
  * Symptomatic congestive heart failure
  * Unstable angina pectoris
  * Cardiac arrhythmia
  * Psychiatric illness or social situation that would limit compliance with study requirements
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No known HIV positivity
* More than 4 weeks since prior radiotherapy
* More than 2 weeks since prior valproic acid
* More than 3 weeks since other prior treatment for AML, including hematopoietic growth factors

  * Hydroxyurea for WBC > 30,000/mm^3 allowed
* Recovered from prior therapy
* No concurrent filgrastim (G-CSF), sargramostim (GM-CSF), epoetin alfa, or darbepoetin alfa
* No other concurrent investigational agents
* No other concurrent anticancer agents or therapies for this cancer

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2006-01; Primary Completion 2009-05 (Actual); Study Completion 2010-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steven Gore, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

REFERENCES:
- [Derived] Schaefer EW, Loaiza-Bonilla A, Juckett M, DiPersio JF, Roy V, Slack J, Wu W, Laumann K, Espinoza-Delgado I, Gore SD; Mayo P2C Phase II Consortium. A phase 2 study of vorinostat in acute myeloid leukemia. Haematologica. 2009 Oct;94(10):1375-82. doi: 10.3324/haematol.2009.009217. PMID 19794082

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 37 participants were enrolled into this trial between January 2006 and August 2007. One patient on Arm A was ineligible; this participant was included in all analyses.
Groups:
- Arm A (Once Daily Vorinostat): Patients receive oral vorinostat (SAHA) once a day on days 1-21. Treatment repeats every 21 days for up to 17 courses in the absence of disease progression or unacceptable toxicity.
- Arm B (Thrice Daily Vorinostat): Patients receive oral SAHA three times a day on days 1-14. Treatment repeats every 21 days for up to 17 courses in the absence of disease progression or unacceptable toxicity.
Period: Overall Study
Arm/Group | Arm A (Once Daily Vorinostat) | Arm B (Thrice Daily Vorinostat)
Started | 15 | 22
Completed | 1 | 4
Not Completed | 14 | 18
Not completed — Death | 3 | 2
Not completed — Adverse Event | 1 | 2
Not completed — Alternative Treatment | 4 | 4
Not completed — Physician Decision | 1 | 1
Not completed — Withdrawal by Subject | 1 | 4
Not completed — Disease Progression | 1 | 3
Not completed — All other reasons | 3 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm A (Once Daily Vorinostat) | Arm B (Thrice Daily Vorinostat) | Total
Number analyzed (Participants) | 15 | 22 | 37
Age, Continuous [Median (Full Range); unit: years] | 67 [41 to 79] | 67 [28 to 81] | 67 [28 to 81]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 5 | 10
  Male | 10 | 17 | 27
Region of Enrollment [Number; unit: participants]
  United States | 15 | 22 | 37
Disease status [Number; unit: participants]
  Relapsed | 12 | 16 | 28
  Untreated | 3 | 6 | 9
AML disease classification [Number; unit: participants]
  Relapsed AML with good risk cytogenetics | 0 | 0 | 0
  All other relapsed AML | 12 | 16 | 28
  Untreated AML patients >= 65 years old | 3 | 3 | 6
  Untreated AML patients with MDS-AML | 0 | 3 | 3
  Untreated AML with >= 3 cytogenetic abnnormalities | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Confirmed Complete Response (CR) Rate
Description: The confirmed complete response rate was estimated by the number of participants with CR divided by the total number of evaluable participants.
  According to the International Working Group (IWG) Criteria for response in AML, to be considered a CR, the following must be met for at least 4 weeks: ANC > 1500/mL, platelets > 100000/mL, no circulating blasts, bone marrow cellularity >20% (biopsy), trilineage maturation, < 5% bone marrow blasts, no auer rods and no extramedullary disease.
Time Frame: Up to 2 years
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Arm A (Once Daily Vorinostat) | Arm B (Thrice Daily Vorinostat)
Number analyzed (Participants) | 15 | 22
percentage of participants | 0 [0 to 23] | 4.5 [0.4 to 24]

2. Secondary Outcome: Time to Progression (TTP)
Description: Time to Progression (TTP) for each patient will be calculated as the number of days from date of registration to either date when disease progression was documented or date of last evaluation without disease progression. The TTP distribution will be estimated using the method of Kaplan-Meier
Time Frame: Duration of study (up to 2 years)
Population: This data was not (and will never be) analyzed. In place of this outcome, time to treatment failure, analyzed and reported as a secondary outcome.
Arm/Group | Arm A (Once Daily Vorinostat) | Arm B (Thrice Daily Vorinostat)
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Overall Survival (OS)
Description: Overall survival (OS) was defined as the time from registration to death of any cause. Surviving patients were censored at the date of last follow-up. The median OS with 95% CI was estimated using the Kaplan Meier method.
Time Frame: Duration of study (up to 2 years)
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Arm A (Once Daily Vorinostat) | Arm B (Thrice Daily Vorinostat)
Number analyzed (Participants) | 15 | 22
days | 105 [55 to 223] | 153 [58 to 229]

4. Secondary Outcome: Number of Participants With Severe (Grade 3, 4 or 5) Adverse Events
Description: Adverse events were graded according to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) version 3.
  Description of Grades:
  Grade 1: Mild Grade 2: Moderate Grade 3: Severe Grade 4: Life-threatening Grade 5: Death
Time Frame: Duration of study (up to 2 years)
Measure: Number; unit: participants
Arm/Group | Arm A (Once Daily Vorinostat) | Arm B (Thrice Daily Vorinostat)
Number analyzed (Participants) | 15 | 22
participants | 10 | 17

5. Other Pre Specified Outcome: Time to Treatment Failure (TTF)
Description: Time to treatment failure (TTF) was defined as the time from registration to until the date of treatment discontinuation of any reason. Patients receiving treatment at the time of analysis were considered censored. The median TTF with 95% CI was estimated using the Kaplan Meier method.
Time Frame: Duration of treatment (up to 17 cycles)
Measure: Median (90% Confidence Interval); unit: days
Arm/Group | Arm A (Once Daily Vorinostat) | Arm B (Thrice Daily Vorinostat)
Number analyzed (Participants) | 15 | 22
days | 42 [26 to 57] | 46 [20 to 71]

ADVERSE EVENTS:
Arm/Group | Arm A (Once Daily Vorinostat) | Arm B (Thrice Daily Vorinostat)
Serious Adverse Events (participants affected / at risk) | 10/15 | 16/22
Other Adverse Events (participants affected / at risk) | 14/15 | 21/22
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A (Once Daily Vorinostat) (N=15) | Arm B (Thrice Daily Vorinostat) (N=22)
Blood disorder (Blood and lymphatic system disorders) | 2 (2) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1) | 3 (3)
Hemoglobin decreased (Blood and lymphatic system disorders) | 0 (0) | 2 (2)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Cecal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 4 (4)
Lower gastrointestinal hemorrhage (Gastrointestinal disorders) | 1 (2) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 3 (3)
Oral hemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Upper gastrointestinal hemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 3 (3)
Chills (General disorders) | 1 (1) | 1 (1)
Death NOS (General disorders) | 1 (1) | 0 (0)
Disease progression (General disorders) | 1 (1) | 0 (0)
Fatigue (General disorders) | 3 (3) | 7 (7)
General symptom (General disorders) | 0 (0) | 1 (1)
Sudden death (General disorders) | 0 (0) | 1 (1)
Catheter related infection (Infections and infestations) | 1 (1) | 1 (1)
Gingival infection (Infections and infestations) | 1 (1) | 0 (0)
Pharyngitis (Infections and infestations) | 0 (0) | 1 (2)
Pneumonia (Infections and infestations) | 1 (1) | 2 (2)
Sepsis (Infections and infestations) | 1 (1) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 2 (2)
Fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Creatine phosphokinase increased (Investigations) | 1 (1) | 0 (0)
Leukocyte count decreased (Investigations) | 0 (0) | 1 (1)
Neutrophil count decreased (Investigations) | 0 (0) | 2 (2)
Platelet count decreased (Investigations) | 1 (1) | 4 (4)
Acidosis (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 2 (3) | 0 (0)
Intracranial hemorrhage (Nervous system disorders) | 1 (1) | 1 (1)
Confusion (Psychiatric disorders) | 0 (0) | 1 (1)
Bronchopulmonary hemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Pharyngeal mucositis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Rash desquamating (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Skin disorder (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Sweating (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Thrombosis (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A (Once Daily Vorinostat) (N=15) | Arm B (Thrice Daily Vorinostat) (N=22)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (2) | 3 (4)
Hemoglobin decreased (Blood and lymphatic system disorders) | 7 (13) | 6 (11)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 2 (3)
Diarrhea (Gastrointestinal disorders) | 3 (4) | 11 (24)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 2 (2)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Ear, nose and throat examination abnormal (Gastrointestinal disorders) | 0 (0) | 1 (1)
Flatulence (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrointestinal disorder (Gastrointestinal disorders) | 0 (0) | 1 (1)
Mucositis oral (Gastrointestinal disorders) | 0 (0) | 2 (2)
Nausea (Gastrointestinal disorders) | 6 (8) | 13 (15)
Stomach pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1) | 7 (7)
Chest pain (General disorders) | 0 (0) | 1 (1)
Edema limbs (General disorders) | 0 (0) | 2 (5)
Fatigue (General disorders) | 12 (22) | 15 (52)
Pain (General disorders) | 0 (0) | 1 (1)
Bladder infection (Infections and infestations) | 0 (0) | 1 (1)
Gingival infection (Infections and infestations) | 1 (1) | 1 (2)
Opportunistic infection (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Sinusitis (Infections and infestations) | 0 (0) | 1 (1)
Radiation recall reaction (dermatologic) (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 1 (1) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 0 (0)
Blood bilirubin increased (Investigations) | 1 (1) | 0 (0)
INR increased (Investigations) | 1 (1) | 0 (0)
Leukocyte count decreased (Investigations) | 6 (10) | 4 (12)
Neutrophil count decreased (Investigations) | 13 (25) | 19 (45)
Platelet count decreased (Investigations) | 14 (28) | 19 (55)
Anorexia (Metabolism and nutrition disorders) | 4 (5) | 9 (19)
Blood glucose increased (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Serum potassium decreased (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (2) | 2 (2)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Ataxia (Nervous system disorders) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 1 (2)
Dysgeusia (Nervous system disorders) | 0 (0) | 2 (2)
Headache (Nervous system disorders) | 0 (0) | 1 (1)
Urinary incontinence (Renal and urinary disorders) | 1 (1) | 0 (0)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 6 (7) | 7 (11)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pharyngeal mucositis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Petechiae (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2)
Rash desquamating (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Sweating (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Hematoma (Vascular disorders) | 0 (0) | 1 (1)
Hemorrhage (Vascular disorders) | 0 (0) | 1 (1)
Hot flashes (Vascular disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less